CLINICAL TRIAL: NCT03425721
Title: Histological and Microbiological Evaluation of Late Occurring Nodules With Hyaluronic Acid Dermal Fillers
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: CMO-US-FAS-0486
Record Dates: First submitted 2018-01-19; First posted 2018-02-08 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Dermal Nodule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All Participants
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention is administered in this study.

SUMMARY:
This study will determine if HA dermal filler late occurring (> 4 weeks and <2 years) nodules are associated with bacterial contamination (independent of filler type) and to characterize the histological response.

ELIGIBILITY:
Inclusion Criteria:

* Have only received HA fillers (no limitation on the brand(s)/product(s) of HA filler used; multiple product use is allowed).
* Present with an unresolved nodule (inflammatory or non-inflammatory) which was first observed > 4 weeks and > 2 years after most recent HA filler treatment and is determined to be greater than 3 millimeters (mm) in diameter by palpation

Exclusion Criteria:

* Have received non-HA fillers (e.g. polyacrylamide, calcium hydroxyapatite, poly-L-lactic acid, polymethylmethacrylate, silicone, expanded polytetrafluoroethylene, collagen) including mixes with HA fillers anywhere in the face.
* Are currently enrolled in a dermal filler clinical trial or previously enrolled in a dermal filler clinical trial with randomized treatment in which the type of dermal filler is unknown (i.e. non-HA filler arm of study).
* Have history of keloid or hypertrophic scarring
* Have received intralesional intervention for the nodule (e.g. hyaluronidase, corticosteroids, antibiotics, 5-fluorouracil).
* Are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who present with late occurring nodules, occurring more than 4 weeks but less than 2 years after the latest injection of any HA soft tissue filler.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2021-04-13 (Actual)

PRIMARY OUTCOMES:
Histological Sampling | 12 Weeks
  Histological lab assessment of biopsy sample for analysis of Hematoxylin and eosin (H&E), orcein, periodic acid-Schiff, gram stain and immunohistochemistry (IHC), with a histopathology assessment to identify possible presence and location of bacteria, mycobacteria, fungus, mold, and/or yeast and the immune/inflammation response within the biopsy.
Microbiological Sampling | 12 Weeks
  Microbiology lab assessment of biopsy sample for analysis of the presence and species of bacteria/mycobacteria within the biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (2):
- United States (2):
  - Skin Care and Laser Physicians (SCLP) of Beverly Hills, West Hollywood, California
  - Assure Surgical, P.C., New York, New York

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Time Frame: For details on when studies are available for sharing, please refer to the link below
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com. For any study not on AllerganClincalTrials.com, please contact IR-CTRegistration.com for assistance. — http://www.AllerganClinicalTrials.com